CLINICAL TRIAL: NCT01490931
Title: Single-dose and Multi-dose Open-label Pilot Trial of the Analgesic Efficacy and Tolerability of Intranasal Ketorolac Tromethamine (SPRIX®) in Dental Implant Surgery Patients With Postoperative Pain.
Brief Title: Intranasal Ketorolac for Postsurgical Pain in Dental Implant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hersh, Elliot V., DMD, MS, PhD (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPRIX IMPLANT 001
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Acute Pain
Keywords: acute pain; dental pain; intranasal ketorolac; dental implant surgery
MeSH Terms: conditions — Acute Pain; Toothache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketorolac nasal spray 31.5 mg (Experimental): Recommended dose according to package insert in 18 - 64 year olds for moderate to moderately severe pain.
  Interventions: Drug: Ketorolac Nasal Spray

INTERVENTIONS:
Drug: Ketorolac Nasal Spray — 15.75 mg nasal spray delivery to each nostril no more than every six hours
  Other Names: SPRIX

SUMMARY:
The surgical placement of dental implants is presently a common procedure performed by oral surgeons, periodontists, and general dentists. The surgery can be performed under local anesthesia and involves the incision of soft tissue to expose the underlying bone, preparation of the implant site using a specialized surgical drill, and.screwing the implant into bone using a specialized headpiece. Dental implant patients experience postoperative pain yet there are no studies in the literature which have evaluated the efficacy of analgesics in this patient population. The current pilot study will evaluate the analgesic effects and tolerability of a recently FDA-approved analgesic formulation of intranasal ketorolac (SPRIX®) in 25 patients who have 1 - 3 dental implants surgically placed. Patients will self administer the ketorolac nasal spray (one spray in each nostril, 31.5 mg total dose) when their postoperative pain reaches at least a moderate severity. Pain intensity and pain relief scores will then be recorded every 20 minutes for the first hour, at 1.5 and 2 hours and then hourly through 6 hours on a validated analgesic diary. Side effects will be recorded when and if they occur. Patients will then transition to a multi-dose phase where they will be allowed to dose with ketorolac as indicated in the package insert (up to 4 times per day for 5 days). Patients will record the time of each dose, a daily assessment of overall efficacy and side effects, and the use of any rescue medication (acetaminophen 650 mg) on a take home diary.

DETAILED DESCRIPTION:
OBJECTIVES

1. Overall Objectives The purpose of this pilot study will be to evaluate the analgesic efficacy and tolerability of intranasal ketorolac employed at doses and dosing intervals stated in the package insert in patients experiencing moderate to severe pain following dental implant surgery. This open label study should provide data that will allow us to estimate sample size for a future placebo-controlled trial in the dental implant surgery population.
2. Primary Outcome Variable(s) To determine if intranasal ketorolac significantly reduces pain intensity scores when compared to baseline pain intensity as measured by the area under the 6-hour pain intensity difference (SPID-6).
3. Secondary Outcome Variable(s) To determine the median onset of first perceptible, confirmed first perceptible, and meaningful pain relief of intranasal ketorolac in dental implant surgery patients.

To compare mean post-dose pain intensity scores at each time-point with the baseline pain intensity score during the initial 6-hour evaluation period.

To calculate the area under the 6-hour pain relief time action curve (TOTPAR-6) for intranasal ketorolac.

To calculate the percentage of subjects who reach a level of at least moderate pain by achieving a score of at least 40 mm on a 100 mm visual analog scale within 5 hours after the completion of surgery.

To determine the mean number of days of analgesic dosing in dental implant surgery patients when employing intranasal ketorolac as their pain medication.

To determine the number of patients taking rescue medication (acetaminophen 650 mg) and the mean number of rescue medication doses taken in dental implant surgery patients when employing intranasal ketorolac as their pain medication.

To determine the overall tolerability of intranasal ketorolac in dental implant surgery patients.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria

1. Male or female between 18 and 64 years of age.
2. Must sign informed consent prior to initiation of any study procedures. The subject must be able to understand and agree to cooperate with study requirements.
3. BMI between 19 and 29 kg/m2.
4. Must require the surgical placement of 1 - 3 dental implants that are being placed in a one or two stage non-immediately loaded surgical procedure employing 2% lidocaine and/or 4% articaine with epinephrine and/or 3% mepivacaine plain for local anesthesia.
5. Females of child-bearing potential must have a negative urine pregnancy test at screening and immediately prior to the initiation of dental implant surgery and must have been using adequate means of birth control (abstinence, oral contraceptive steroids, intrauterine device (IUD), etc.) for at least one month prior to study entry and during the study.
6. In the opinion of the investigators the subject can safely tolerate ketorolac and acetaminophen.

   -

Exclusion Criteria:

Key Exclusion Criteria

1. Require the placement of more than 3 implants or require extensive bone grafting in addition to implant placement.
2. Need to administer anxiolytic/sedation drugs during surgery other than nitrous oxide/oxygen.
3. Need to administer the long acting local anesthetic bupivacaine with 1:200,000 epinephrine.
4. Implant(s) that are going to be immediately loaded on the day of surgery
5. Females that are pregnant or breast feeding
6. Allergies or hypersensitivity (aspirin sensitive asthma) to ketorolac, aspirin, ibuprofen, other NSAIDs, or acetaminophen.
7. History of gastrointestinal ulcers and/or bleeding.
8. On warfarin, dicumarol, clopidogrel or any other anticoagulant or antiplatelet therapy other than low dose (81 mg - 325 mg) aspirin.
9. Clinically significant kidney or liver disease where the intake of NSAIDs or acetaminophen would put the subject at undo risk.
10. Blood pressure greater than 160/95 at the time of screening or immediately before surgery.
11. Inflammation of the nasal mucosa or upper respiratory tract infection
12. Have ingested any analgesic agent within 48 hours of surgery.

    -

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot V Hersh, DMD, MS, PhD, Principal Investigator — Univeristy of Pennsylvania School of Dental Medicine
Locations (1):
- University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Al-Khabbaz AK, Griffin TJ, Al-Shammari KF. Assessment of pain associated with the surgical placement of dental implants. J Periodontol. 2007 Feb;78(2):239-46. doi: 10.1902/jop.2007.060032. PMID 17274712
- [Background] Hersh EV, Levin LM, Adamson D, Christensen S, Kiersch TA, Noveck R, Watson G 2nd, Lyon JA. Dose-ranging analgesic study of Prosorb diclofenac potassium in postsurgical dental pain. Clin Ther. 2004 Aug;26(8):1215-27. doi: 10.1016/s0149-2918(04)80033-x. PMID 15476903
- [Result] Bockow R, Korostoff J, Pinto A, Hutcheson M, Secreto SA, Bodner L, Hersh EV. Characterization and treatment of postsurgical dental implant pain employing intranasal ketorolac. Compend Contin Educ Dent. 2013 Sep;34(8):570-6. PMID 24564610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients in PENN periodontal clinic or faculty practice requiring 1 to 3 dental implants employing lidocaine with epinephrine for anesthesia without significant bone augmentation
Pre-assignment Details: Subjects not experiencing moderate pain (at least 40 mm on the pain intensity VAS and moderate or severe pain on the 4-point categorical scale) within 4 hours of surgery were not dosed with ketorolac. Of the 28 enrolled subjects, 25 (89%) achieved at least moderate pain and were dosed.
Groups:
- Ketorolac Nasal Spray 31.5 mg (SPRIX): Recommended dose according to package insert in 18 - 64 year olds for moderate to moderately severe pain.
  Ketorolac Tromethamine Nasal Spray: 15.75 mg nasal spray delivery to each nostril no more than every six hours
Period: Overall Study
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pilot Study. No power analysis performed.
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 25
pain intensity on 100 mm visual analog scale (VAS). 0=No pain 100=worst possible pain [Mean (Standard Deviation); unit: units on a scale] | 54.4 (14.3)

OUTCOME MEASURES:

1. Secondary Outcome: The Median Onset of First Perceptible Pain Relief of Intranasal Ketorolac in Dental Implant Surgery Patients
Description: Data will be obtained employing the well-described double stop watch technique
Time Frame: Censored at 6 hours
Measure: Median (95% Confidence Interval); unit: seconds
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
seconds | 86 [64 to 172]

2. Primary Outcome: Comparison of Pain Intensity Scores at 20 Minutes With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period.
Description: Pain intensity scores will be recorded by patient employing a standard 100 mm visual analog scale
Time Frame: 20 minutes post dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 14.3 (4.1)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); Changes in pain intensity on the VAS were statistically compared to baseline pain utilizing paired t tests with Bonferroni corrections for multiple comparisons. The median onsets of first perceptible and meaningful relief (with 95% confidence intervals) were calculated and then used to construct Kaplan-Meier Curves of the distribution of pain relief times; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P value adjusted with Bonferroni corrections for multiple comparisons

3. Secondary Outcome: Percentage of Subjects Who Reach a Level of at Least Moderate Pain by Achieving a Score of at Least 40 mm on a 100 mm Visual Analog Scale Within 5 Hours After the Completion of Surgery.
Time Frame: Up to 5 hours after last suture is placed
Population: All subjects (regardless of pain intensity) receiving one to three dental implants
Measure: Number; unit: percentage of participants
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 28
percentage of participants | 89

4. Secondary Outcome: Most Frequent Number of Days of Analgesic Dosing in Dental Implant Surgery Patients When Employing Intranasal Ketorolac as Their Pain Medication.
Description: Self explanatory
Time Frame: Up to 5 days
Measure: Number; unit: days
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
days | 3

5. Secondary Outcome: Median Onset of Meaningful Pain Relief
Description: Measure obtained using recognized double-stop watch technique. Patient is asked to depress the second stop watch when pain relief is meaningful to them. Each patient decides what meaningful relief is for them.
Time Frame: At time of depressing meaningful relief stopwatch up to 6 hours.
Measure: Median (95% Confidence Interval); unit: seconds
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
seconds | 172 [132 to 735]

6. Primary Outcome: Comparison of Pain Intensity Scores at 40 Minutes With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period.
Description: VAS pain intensity score at 40 minutes post-dose
Time Frame: 40 minutes post dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 10.1 (2.2)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

7. Primary Outcome: Comparison of Pain Intensity Scores at 60 Minutes With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period
Description: VAS pain intensity score 60 minutes after dosing.
Time Frame: 60 minutes post dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 10.6 (1.8)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

8. Primary Outcome: Comparison of Pain Intensity Scores at 90 Minutes With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period
Time Frame: 90 minutes post-dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 9.6 (2.2)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

9. Primary Outcome: Comparison of Pain Intensity Scores at 2 Hours With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period
Time Frame: 2 Hours
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 9.1 (2.0)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

10. Primary Outcome: Comparison of Pain Intensity Scores at 3 Hours With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period
Time Frame: 3 hours post-dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 9.6 (2.2)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0001, t-test, 2 sided

11. Primary Outcome: Comparison of Pain Intensity Scores at 4 Hours With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period
Time Frame: 4 Hours post-dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 10.0 (2.0)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

12. Primary Outcome: Comparison of Pain Intensity Scores at 5 Hours With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period
Time Frame: 5 Hours post-dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 16.2 (4.3)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

13. Primary Outcome: Comparison of Pain Intensity Scores at 6 Hours With the Baseline Pain Intensity Score During the Initial 6-hour Evaluation Period
Time Frame: 6 Hours post-dose
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Number analyzed (Participants) | 25
millimeters | 19.8 (3.7)
Statistical Analysis 1: Comparison: Ketorolac Nasal Spray 31.5 mg (SPRIX); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Ketorolac Nasal Spray 31.5 mg (SPRIX)
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 14/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Nasal Spray 31.5 mg (SPRIX) (N=25)
Nasal burning or stinging (Respiratory, thoracic and mediastinal disorders) | 9 (9) — Transient nasal burning on dosing in 9/25 (36%) of subjects
Throat burning (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Transient throat burning on dosing 3/25 subjects (12%)
Headache (Nervous system disorders) | 3 (3) — 3 of 25 (12%) reported headache sometime during 5 day evaluation period
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Sneezing on dosing 2/25 (8%)
Constipation (Gastrointestinal disorders) | 1 (1)
Difficulty breathing sensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Transient difficulty breathing sensation immediately after dosing
Ears popping sensation (Ear and labyrinth disorders) | 1 (1) — Transient immediately after dosing
Perspiring (Skin and subcutaneous tissue disorders) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Watery eyes (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The major weakness of this study was its open-label design and lack of a placebo control and an active comparator drug. The study was also not powered to determine differences between the sites of implant placement and the number of implants placed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes